CLINICAL TRIAL: NCT03139188
Title: Palliative Care Transfer Announcements: Qualitative Analysis of the Perspective of Physicians and Their Patients With Cancer
Brief Title: Palliative Care Unit Transfert Announcements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6789
Record Dates: First submitted 2017-04-21; First posted 2017-05-03 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: Cancer; incurable pathologies; palliative care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The course of care of a patient with a cancer whose evolution is pejorative, is marked by difficult announcements, called "bad news". In the palliative phase, prognostic announcements are at the forefront. Of these, the announcement of a transfer to the Palliative Care Unit has not been the subject of any specific studies to the best of our knowledge. It therefore seemed interesting to us to explore the stakes of this particular announcement, a source of upheaval for the doctor and the patient, by gathering the point of view of each one.

The objective of our study is to analyze the methods of announcing a transfer to the Palliative Care Unit and the perception of this announcement by the doctor and his patient with an incurable cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with solid cancer or malignant haemopathy in palliative phase transferred from a HUS service to the HUS UnASP and informed of this transfer by the originating doctor .

HUS senior hospital doctors, supporting patients with solid cancers or malignant hemopathies.

Exclusion Criteria:

* Patients whose clinical state does not allow for maintenance (tiredness, confusion) or difficult communication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with solid cancer or malignant haemopathy in palliative phase transferred from a HUS service to the HUS UnASP
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Analysis of semi-structured interviews exploring how the physician analyzes and feels the announcement of the transfer to the Palliative Care Unit and how the patient receives and disseminates this information | 72 hours after the transfer of the patient the to the Palliative Care Unit

CONTACTS AND LOCATIONS:
Overall Officials: Virginie LEROY, MD, Study Director — University Hospital, Strasbourg, France; Laurent CALVEL, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service : Unité de soins d'Accompagnement de soins de Support et de soins Palliatifs (UnASP), Strasbourg, France

IPD SHARING:
Plan to Share IPD: No